CLINICAL TRIAL: NCT03025230
Title: Effectiveness of Dry Needling and Intramuscular Electrostimulation in the Treatment of Myofascial Trigger Points in Patients With Neck Pain
Brief Title: Dry Needling Versus Intramuscular Stimulation in the Management of the Myofascial Trigger Points
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alcala (Other)
Responsible Party: Principal Investigator, Prof. Dr. Daniel Pecos Martín, Dr. Pecos-Martin, Daniel (Principal Investigator), University of Alcala
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: M2012119/20130409
Record Dates: First submitted 2017-01-16; First posted 2017-01-19 (Estimated); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Trigger Point Pain, Myofascial; Muscle Pain; Myofascial Pain Syndrome
MeSH Terms: conditions — Myofascial Pain Syndromes; Myalgia | interventions — Dry Needling; Electric Stimulation

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Dry needling technique and the application of a rectangular, biphasic, asymmetric analgesic electric current by selecting a frequency of 2 Hz with a pulse width 40 μs, with an intensity located at the tolerance threshold and for a time of 20 minutes.
  Interventions: Other: Dry needling and electric stimulation
- Control group (Active Comparator): Dry technique in PG.The needle will be moved in-and-out into different directions to encounter sensitive spots in PG region.
  Interventions: Other: Dry needling

INTERVENTIONS:
Other: Dry needling and electric stimulation — Dry needling technique and the application of electric stimulation of levator scapulae PG
  Arms: Experimental group
Other: Dry needling — Treatment of PG with a filiform needle in levator scapulae muscle
  Arms: Control group

SUMMARY:
Hypothesis The application of intramuscular electrostimulation will be more effectiveness than the dry needling in myofascial trigger points treatment.

Objetives:

To determine the effectiveness of intramuscular electrostimulation in the treatment of trigger points of the levator scapula muscle for the improvement of pain in mechanical cervicalgia.

Participants: Subjects with diagnosed of myofascial pain syndrome in cervical region and active trigger points in levator scapulae muscle, randomly assigned to experimental or control group.

Intervention: Control group: one session of dry needling in active trigger points; experimental group: one session of intramuscular stimulation in active trigger points.

Main Outcomes Measures: Pain, pressure pain threshold (PPT), active cervical range of motion and strength muscle . The measures will be taken before, after and one week after the interventions.

DETAILED DESCRIPTION:
The muscle pain is one of the most common forms of musculoskeletal pain. Within muscular pain, the presence of myofascial trigger points (PG) in the musculature is a important and prevalent problem.

Currently one the techniques most used in the treatment of PG is dry needling. Dry needling has been shown effective in the treatment of neck pain associated with PGs.

To our knowledge, there are no studies that they have compared the effectiveness of dry needling and intramuscular stimulation by applying an electric current.

This study is a randomized clinical trial that aims to demonstrate that the application of an electric current associated with dry needling in the treatment of PG.

In this study we will treat subjects with cervical pain who they have active PGs in the levator scapulae muscle.

ELIGIBILITY:
Inclusion Criteria:

* Cervical pain.
* Active trigger points in levator scapulae muscle

Exclusion Criteria:

* Pain Irradiation toward upper limb
* Psychological disorders
* Whiplash.
* Neuropathic symptoms
* Cervical and / or Shoulder Spine Surgery

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Pressure Pain Threshold (PPT) | Change from baseline at one week
  An algometer Wagner FPI 10-WA will be used to determine the PPT in levator scapulae trigger points

SECONDARY OUTCOMES:
Pain Visual Analogue Scale | Change from baseline at one week
  The pain VAS is a unidimensional measure of pain intensity, which has been widely used in diverse adult populations. The VAS is a straight horizontal line of fixed length, usually 100 mm. The ends are defined as the extreme limits of the parameter to be measured from 0 (no pain) to 10 (maximum pain). All the subjects will showed their pain level.
Strength in cervical latero-flexion | Change from baseline at one week
  Dynamic dynamometry with MicroFet-2 will be used while patients will positioned in seated. From this position, patients will performed lateral - flexion

CONTACTS AND LOCATIONS:
Overall Officials: Tomás Gallego-Izquierdo, Doctor, Study Director — Alcala University
Locations (1):
- Patricia Martínez Merinero, Alcalá de Henares, Madrid, Spain